CLINICAL TRIAL: NCT07048899
Title: Effects of Irrisept Irrigation in Emergency General Surgery Cases on SSI Rates
Brief Title: Irrisept in Emergency General Surgery Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Principal Investigator, Brittany Wagner, General Surgery Resident, The University of Texas Health Science Center at Tyler
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-122
Record Dates: First submitted 2025-06-11; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Emergency Surgery; Surgical Site Infections
Keywords: Irrisept; Surgical Irrigation; Surgical Site Infection; Emergency General Surgery; Acute Care Surgery; Normal Saline Irrigation
MeSH Terms: conditions — Surgical Wound Infection | interventions — Chlorhexidine; Saline Solution; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Normal Saline) (Placebo Comparator): Irrigation with Normal Saline
  Interventions: Drug: Normal Saline
- Intervention (Irrisept) (Experimental): Irrigation with Irrisept
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — Intraperitoneal irrigation with Irrisept solution
  Other Names: Irrisept
  Arms: Intervention (Irrisept)
Drug: Normal Saline — Intraperitoneal irrigation with normal saline
  Other Names: Standard of Care
  Arms: Standard of Care (Normal Saline)

SUMMARY:
This is a single institution, randomized study conducted to determine if irrigation with Irrisept in emergency general surgery patients results in lower surgical site infections compared to normal saline irrigation.

ELIGIBILITY:
Inclusion Criteria:

* All patients (>18 years old at time of enrollment) who are hospitalized at UT Tyler and undergo an open (or conversion to open) wound class 2-4 surgical procedure for an emergent surgical condition.

Exclusion Criteria:

* Those <18 years of age
* Pressure wounds
* Superficial abscesses (as primary diagnosis)
* intra-abdominal abscess due to previous technical failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | Time of enrollment to 30 days
  Determine if the rate of SSI is different

SECONDARY OUTCOMES:
Length of Stay | From date of admission until date of discharge from the hospital, assessed up to 30 days post-operatively
  Number of days admitted to hospital
Incidence of SSI and surgical wound class with the use of Irrisept | Time of enrollment to 30 days
  Correlation between surgical wound class and the use of Irrisept on the incidence of SSI
Readmission Rates due to SSI | From day of surgery to 30 days
  How often a patient has to be re-admitted to the hospital for a surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the result publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning after completion of project and ending 5 years after publication of results